CLINICAL TRIAL: NCT00906438
Title: Effects of 2006-RD-05 on Salivary and Serum IgA Levels in Healthy Subjects
Brief Title: Effects of 2006-RD-05 on Salivary and Serum Immunoglobulin A (IgA) Levels in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: innoVactiv Inc. (Industry)
Responsible Party: Scientific Director, Health & Nutrition, innoVactiv inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2006-RD-05-CLN1
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Treated (Experimental)
  Interventions: Dietary Supplement: 2006-RD-05

INTERVENTIONS:
Dietary Supplement: 2006-RD-05 — 300 mg daily, once a day for 28 consecutive days
  Arms: Treated
Dietary Supplement: Placebo — Capsule similar in shape, weight and color from active, once a day for 28 consecutive days
  Arms: Control

SUMMARY:
It is already known from animal studies that the study drug can improve mucosal immunity as shown by increased serum and mucosal IgA secretion. This study will evaluate the safety of an oral intake of the natural product 2006-RD-05 at the recommended daily dose of 300 mg. In addition, this trial will aim to determine if this intake is able ot improve serum and salivary IgA synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 - 60
* In good health
* BMI between 20 and 30 kg/m2
* Non-smoking

Exclusion Criteria:

* Allergic to study drug
* Use of immune-modulating drugs
* Uncontrolled hypertension (Systolic > 140 or diastolic > 90)
* Women of childbearing age not using proper contraception, that is pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | Baseline, 14 days, 28 days

SECONDARY OUTCOMES:
Serum IgA titers | Baseline, 14 days, 28 days
Salivary IgA titers | Baseline, 14 days, 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institut des Nutraceutiques et des Aliments Fonctionnels (INAF), Québec, Quebec, Canada